CLINICAL TRIAL: NCT02924051
Title: Interventions in Nutrition Education and Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frances Hardin-Fanning, PhD, RN (Other)
Responsible Party: Sponsor-Investigator, Frances Hardin-Fanning, PhD, RN, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14-0020-P2H
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-05

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Control/Intervention Groups (3 sites in each group)
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Motivational Interview (MI) (Experimental): Intervention group participants receive cooking skills and nutritional education via cookbooks, cooking classes, food preparation tools and prepared food dishes to take home to their families, along with monthly motivational interviewing conducted by a trained registered nurse
  Interventions: Behavioral: Motivational Interviewing
- Cooking Skills/Nutritional Education (Active Comparator): Participants in this arm receive cooking skills and nutritional education via cookbooks, cooking classes, food preparation tools and prepared food dishes to take home to their families.
  Interventions: Behavioral: Cooking skills and nutritional education

INTERVENTIONS:
Behavioral: Motivational Interviewing — Baseline and monthly assessment of barriers/facilitators of dietary change, ambivalence to change and "coaching" to resolve barriers and ambivalence.
  Arms: Motivational Interview (MI)
Behavioral: Cooking skills and nutritional education — Participants in this group will develop an understanding of healthy food options and healthy food preparation.
  Arms: Cooking Skills/Nutritional Education

SUMMARY:
Healthy eating can be difficult for people who live in poor, geographically isolated regions of the United States. In particular, people who live in Appalachia often experience food insecurity (i.e., their access to adequate food is limited by a lack of money and other resources at times during the year) and lack of access to healthy foods. This pilot study evaluates the effectiveness of motivational interviewing in helping individuals who live in these austere regions improve their diets in the context of limited resources and healthy food availability

DETAILED DESCRIPTION:
Participants in three of the counties will receive an education/skills intervention paired with a form of coaching called motivational interviewing (MI) conducted by a trained registered nurse. Three similar counties that do not border any of the intervention counties are serving as controls (these counties receive the same nutrition education/skills intervention without motivational interviewing). All participants will receive cookbooks, cooking classes, food preparation tools, and prepared food dishes to take home to their families. The investigators will measure the impact of motivational interviewing on fresh fruit and vegetable consumption, saturated fat consumption and number of meals cooked at home.

ELIGIBILITY:
Inclusion Criteria:

• People who live in one of six rural Kentucky food desert counties

Exclusion Criteria:

* <16 years old
* Unable to read/write English
* Any GI malabsorption disorder that prevents high fiber consumption

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
Data being compiled
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Will be available upon request June 30, 2018 (following publication/presentation of primary/secondary outcome results). Data will be available for 6 years.
Access Criteria: Data, free of identifiers, will be provided in Excel spreadsheets to requesting researchers to the PI via email (fdbowe2@uky.edu) after June 30, 2018. Both the University of Kentucky Medical IRB and Data Safety Monitoring Board will be asked to review the request prior to release. Researchers must state purpose of the request, intent of data analysis, and acknowledge the PI in subsequent publications/presentations by signing the University of Ky College of Nursing Data Use Agreement and Letter of Intent.

RESULTS

PARTICIPANT FLOW:
Groups:
- Cooking Skills/Nutrition Education: Control group received cookbooks, cooking classes, food preparation tools and prepared food dishes to take home to their families.
- Cooking Skills/Nutrition Education/Motivational Interviewing: Intervention group participants received cookbooks, cooking classes, food preparation tools and prepared food dishes to take home to their families, along with monthly motivational interviewing conducted by a trained registered nurse.
  Motivational Interviewing: Baseline and monthly assessment of barriers/facilitators of dietary change, ambivalence to change and "coaching" to resolve barriers and ambivalence.
Period: Overall Study
Arm/Group | Cooking Skills/Nutrition Education | Cooking Skills/Nutrition Education/Motivational Interviewing
Started | 82 | 106
Completed | 81 | 97
Not Completed | 1 | 9
Not completed — Withdrawal by Subject | 1 | 9

BASELINE CHARACTERISTICS:
Groups:
- Control: Control group received cookbooks, cooking classes, food preparation tools and prepared food dishes to take home to families.
- Intervention: Intervention group participants received cookbooks, cooking classes, food preparation tools and prepared food dishes to take home to their families, along with monthly motivational interviewing conducted by a trained registered nurse.
  Motivational Interviewing: Baseline and monthly assessment of barriers/facilitators of dietary change, ambivalence to change and "coaching" to resolve barriers and ambivalence.
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 82 | 106 | 188
Age, Continuous [Mean (Full Range); unit: years] | 55.4 [16 to 81] | 50.3 [19 to 76] | 54.9 [16 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 99 | 176
  Male | 5 | 7 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 1 | 3
  White | 79 | 104 | 183
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 82 | 106 | 188

OUTCOME MEASURES:

1. Primary Outcome: Change in BLOCK Fruit/Vegetable/Fiber Screener From Baseline at 12 Months
Description: Block Fruit/Vegetable/Fiber Screener is a tool that ranks usual intake of fruit, vegetables, and fiber. Total fruit/vegetable/fiber score can range from 0-50 with higher numbers reflecting greater frequency of fruit, vegetable and fiber consumption.
Time Frame: Baseline, 12 months
Population: Participants who completed the Block Screener at baseline and post-intervention (12 months)
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Cooking Skills/Nutrition Education: Control group received cookbooks, cooking classes, food preparation tools and prepared food dishes to take home to families.
Arm/Group | Cooking Skills/Nutrition Education | Cooking Skills/Nutrition Education/Motivational Interviewing
Number analyzed (Participants) | 54 | 60
units on a scale
  Baseline | 16.6 [2 to 34] | 15.9 [5 to 30]
  12 months | 18.0 [6 to 35] | 16.3 [6 to 29]
Statistical Analysis 1: Comparison: Cooking Skills/Nutrition Education vs Cooking Skills/Nutrition Education/Motivational Interviewing; Test type: Equivalence — With an alpha level of .05 and effective (post-attrition) sample size of approximately 25 participants per county, and 3 counties per treatment group, the power of the group comparison was at least 80%, assuming an ICC of .01 or less, and an observed difference in proportions of .25. The anticipated power for the longitudinal comparison of continuous outcomes was expected to be even greater under these assumptions given the greater power for the parametric tests; p = 0.26, t-test, 2 sided; Mean Difference (Final Values) = 1.12

2. Secondary Outcome: Average Saturated Fatty Acid Intake/Day
Description: Using the NCI DHQ II, respondents' frequency of consumption of foods (i.e., meats and oils) and portion size, dietary saturated fat consumption was calculated as average grams/day. Higher grams/day reflect higher consumption of saturated fatty acids.
Time Frame: Baseline, 12 months
Population: Number of participants completing the NCI DHQ II survey
Measure: Mean (Standard Deviation); unit: grams/day
Groups:
- Cooking Skills/Nutrition Education: Participants in the control group received cookbooks, cooking classes, food preparation tools and prepared food dishes to take home to their families.
  Motivational Interviewing: Baseline and monthly assessment of barriers/facilitators of dietary change, ambivalence to change and "coaching" to resolve barriers and ambivalence.
Arm/Group | Cooking Skills/Nutrition Education | Cooking Skills/Nutrition Education/Motivational Interviewing
Number analyzed (Participants) | 32 | 36
grams/day
  Baseline | 26.8 (15.4) | 23.8 (14.3)
  Post-Intervention (12 mos) | 19.2 (9.6) | 21.6 (17.9)

3. Secondary Outcome: Frequency of Fast Food Consumption
Description: Fast food consumption was measured using a single item on the National Cancer Institute Diety History Questionaire (NCI DHQ II) "How often did you eat beef hamburgers or cheeseburgers from a fast food or other restaurant?" Responses are selected from 11 pre-determined options increasing in frequency from "never" to "2 or more times per day." Values range from 0 to 10; higher values indicate an increased frequency of fast food consumption.
Time Frame: Baseline and 12 months
Population: Participants completing the NCI DHQ II question related fast food comsumpsion
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Cooking Skills/Nutrition Education/MI: Intervention group participants received cookbooks, cooking classes, food preparation tools and prepared food dishes to take home to their families, along with monthly motivational interviewing conducted by a trained registered nurse.
  Motivational Interviewing: Baseline and monthly assessment of barriers/facilitators of dietary change, ambivalence to change and "coaching" to resolve barriers and ambivalence.
Arm/Group | Cooking Skills/Nutrition Education | Cooking Skills/Nutrition Education/MI
Number analyzed (Participants) | 27 | 38
units on a scale
  Baseline | 3.56 (.49) | 3.16 (0.53)
  12 months | 3.78 (0.50) | 3.03 (0.46)
Statistical Analysis 1: Comparison: Cooking Skills/Nutrition Education/MI; Comparison of Cooking Skills/Nutrition Education/MI at baseline and 12 months; Test type: Superiority; p = 0.36, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Adverse event data were monitored over the entire 12 month period of the study. No adverse or serious adverse events were reported in this study.
Description: Adverse event monitoring was based on Clinical Trials definitions.
Groups:
- Control: Control group received cookbooks, cooking classes, food preparation tools and prepared food dishes to take home to their families.
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/106
Other Adverse Events (participants affected / at risk) | 0/82 | 0/106

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No